CLINICAL TRIAL: NCT01259258
Title: Dye Assisted Lymphatic Sparing Varicocelectomy,Prospective Randomized Study
Brief Title: Dye Assisted Lymphatic Sparing Subinguinal Varicocelectomy
Acronym: varicocele
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: mohamed el ayed, masoura university
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: varicocele
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-11

CONDITIONS: Varicocele
Keywords: varicocele, methylene blue, varicocelectomy, hydrocele,
MeSH Terms: conditions — Varicocele; Testicular Hydrocele

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varicocelectomy with dye (Active Comparator): subinguinal varicocelectomy for 40 patients who received 2 ml intratunical space injection of methylene blue before spermatic vein ligation
  Interventions: Procedure: without dye varicocelectomy
- without dye varicocelectomy (Active Comparator): 40 controls in whom no mapping technique was adopted in the period between
  Interventions: Procedure: without dye varicocelectomy

INTERVENTIONS:
Procedure: without dye varicocelectomy — 40 controls in whom no mapping technique was adopted in the period between
  Other Names: optical subinguinal varicocelectomy
  Arms: varicocelectomy with dye
Procedure: without dye varicocelectomy — 40 controls in whom no mapping technique was adopted in the period between
  Other Names: microoptic subinguinal varicocelectomy
  Arms: without dye varicocelectomy

SUMMARY:
We prospectively compared outcomes of subinguinal varicocelectomy for 40 patients who received 2 ml intratunical space injection of methylene blue before spermatic vein ligation with 40 controls in whom no mapping technique was adopted in the period between January 2008 and Feb. 2010, in Mansoura university hospital ward 7.After surgery, the patients were assessed at 2 weeks,6 and 12 months for varicocele recurrence, hydrocele formation, atrophy, pain or other complications with mean follow up was 15+ 7months.

DETAILED DESCRIPTION:
Methods. We prospectively compared outcomes of subinguinal varicocelectomy for 40 patients who received 2 ml intratunical space injection of methylene blue before spermatic vein ligation with 40 controls in whom no mapping technique was adopted in the period between January 2008 and Feb. 2010, in Mansoura university hospital ward 7.After surgery, the patients were assessed at 2 weeks,6 and 12 months for varicocele recurrence, hydrocele formation, atrophy, pain or other complications with mean follow up was 15+ 7months.

Results: There were no intraoperative complications in either group. There were no adverse reactions, scrotal haematomas or atrophy. In group 1, no patient had a hydrocele at 3 months after surgery. By contrast, in group 2 (surgery alone) there were four cases of secondary hydrocele (10%; P=0.025)); no testicular hypertrophy was observed following lymphatic sparing surgery , One patient in each group had varicocele recurrence. Pregnancy was reported in 30 patients (37.5%) during a follow up period, 17 of them (42.5%) were group(1),P >0.34. difference was not significantly different among the two groups

ELIGIBILITY:
Inclusion Criteria:

* all left sided varicocele with impaired sperm counts, testicular pain and/or testicular atrophy

Exclusion Criteria:

* were preexisting hydrocele, previous groin surgery, concomitant hernia, allergy against methylene blue

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
postoperative complication | 30 days
  hydrocele

SECONDARY OUTCOMES:
recurrence, pregnancy, semen parameter | one year
  recurrence, pregnancy, semen parameter

CONTACTS AND LOCATIONS:
Overall Officials: ayman elnakeeb, MD, Study Chair — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Background] Ghanem H, Anis T, El-Nashar A, Shamloul R. Subinguinal microvaricocelectomy versus retroperitoneal varicocelectomy: comparative study of complications and surgical outcome. Urology. 2004 Nov;64(5):1005-9. doi: 10.1016/j.urology.2004.06.060. PMID 15533495
- [Background] Zini A, Fischer A, Bellack D, Noss M, Kamal K, Chow V, Mak V. Technical modification of microsurgical varicocelectomy can reduce operating time. Urology. 2006 Apr;67(4):803-6. doi: 10.1016/j.urology.2005.10.044. Epub 2006 Mar 29. PMID 16566968
- [Background] Schwentner C, Oswald J, Lunacek A, Deibl M, Bartsch G, Radmayr C. Optimizing the outcome of microsurgical subinguinal varicocelectomy using isosulfan blue: a prospective randomized trial. J Urol. 2006 Mar;175(3 Pt 1):1049-52. doi: 10.1016/S0022-5347(05)00410-6. PMID 16469616
- [Background] Atteya A, Amer M, AbdelHady A, Al-Azzizi H, Ismael E, Abdel-Gabbar M, Shamloul R. Lymphatic vessel hydrodissection during varicocelectomy. Urology. 2007 Jul;70(1):165-7. doi: 10.1016/j.urology.2007.04.012. PMID 17656230
- [Derived] Abd Ellatif ME, El Nakeeb A, Shoma AM, Abbas AE, Askar W, Noman N. Dye assisted lymphatic sparing subinguinal varicocelectomy. A prospective randomized study. Int J Surg. 2011;9(8):626-31. doi: 10.1016/j.ijsu.2011.07.430. Epub 2011 Aug 23. PMID 21875697
- See also: mansoura university — http://www.mans.edu.eg/